CLINICAL TRIAL: NCT01117389
Title: Human Papillomavirus (HPV) Vaccination Among Survivors of Childhood Cancer
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Other Study IDs: HPV1
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Human Papillomavirus
Keywords: Human Papillomavirus Vaccination; Childhood cancer survivors; cervical cancer; sexually transmitted infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mothers of Childhood cancer survivors: Mothers or female primary caregivers of active patients (aged 9-17) and young adult female patients aged 18-26 in the After Completion of Therapy (ACT) clinic at SJCRH. Mothers or female primary caregivers of active patients (aged 9-17) and young adult female patients aged 18-26 in the ACT clinic surviving childhood cancer will be asked to complete a questionnaire which queries sociodemographic, medical, and psychological variables which may relate to HPV vaccination.
- Acquaintance control Group: Mothers or female primary caregivers ( with daughters aged 9-17) and young adult females aged 18-26 referred for study participation by participants from the ACT clinic. Participants have daughters aged 9-17 years or young adult females aged 18-26 at the time of study enrollment For those acquaintance controls electing to complete the paper-and-pencil questionnaire, the study team will send it to them in the mail along with a pre-addressed, stamped, return envelope. For those electing to complete the on-line questionnaire, the participant's email address will be collected and a secured link to our on-line questionnaire will be sent to them in an email.
  A supplemental community control sample (meeting the inclusion and exclusion criteria outlined above) will also be utilized via the subject pool in the Department of Psychology at The University of Memphis.

SUMMARY:
This study will focus on the primary objectives:

* To estimate the prevalence of HPV vaccination among a large cohort of childhood cancer survivors and an acquaintance control group.
* To describe the difference in HPV vaccination rate and HPV vaccination intent among preadolescent/adolescent females surviving childhood cancer and an acquaintance control group.

This study will also focus on the secondary objectives:

* To examine sociodemographic, medical, and psychological differences between those who have/have not initiated HPV vaccination and between those who do/do not intend to get vaccinated in the future.
* To assess the general predictive influence of sociodemographic, medical, and psychological variables on HPV vaccination and intent among mothers with preadolescent/adolescent daughters.

DETAILED DESCRIPTION:
Effective vaccination is now available to prevent human papillomavirus (HPV), the most common sexually transmitted infection and the cause of cervical cancer, the second most common cancer among women worldwide. HPV vaccine uptake is particularly important for females surviving childhood cancer, many of whom are at high risk for HPV complications due to the direct and indirect effects of cancer treatment. Thus, Version 3.0 of the Children's Oncology Group Long-Term Follow-Up Guidelines for Survivors of Childhood, Adolescent and Young Adult Cancer has recently recommended HPV vaccination for all eligible females surviving childhood cancer. Because this vaccine was only FDA approved in 2006, little is known about the complexity of vaccination uptake among those surviving cancer, and how the factors influencing vaccination decision-making differ among families with and without a history of pediatric cancer.

The purpose of this exploratory study is to estimate the prevalence of HPV vaccination and to assess predictors of HPV vaccination (and intent) among 9-26 year old females who have survived childhood cancer, while making comparisons to healthy acquaintance controls. In a cross-sectional design, those surviving childhood cancer (and acquaintance controls) will be asked to complete a questionnaire which queries sociodemographic, medical, and psychological variables which may relate to HPV vaccination or intent. Current vaccination rates will be examined and factors which associate with HPV vaccination (and intent) will be identified. Findings of the present study will inform recruitment strategies for future studies examining the immunogenicity, safety, tolerability, and behavioral outcomes of HPV vaccination among females surviving childhood cancer. More immediately, this work will further our understanding of familial decision-making regarding HPV vaccination among female survivors of childhood cancer and will determine whether vaccination recruitment models developed for healthy adolescents and young adults generalize to the pediatric cancer population.

ELIGIBILITY:
Inclusion Criteria- Mothers of ACT patients

1. Active females patients (aged 18-26 years) or mothers/female primary caregivers of minor female patients (aged 9-17 years) in the After Completion of Therapy (ACT) clinic at St. Jude Children's Research Hospital (SJCRH).
2. Proficient in reading and writing English.
3. Cognitively intact such that the study questionnaire can be understood and completed.
4. Participant is willing and able to provide informed consent according to institutional guidelines.

Inclusion criteria for acquaintance control participants:

An acquaintance control sample will be comprised of a community sample of adult women (aged 18-26 years) and mothers with daughters in the 9-17 year age range who are acquainted with the ACT patient's family.The primary feature distinguishing the acquaintance controls from the SJCRH sample is the presence/nonpresence of personal (for controls aged 18-26) or daughter's (for maternal controls) cancer history.

The following represents the inclusion criteria for acquaintance control participants:

1. Females (aged 18-26 years) or mothers/female primary caregivers (with daughters aged 9-17 years) referred for study participation by adult survivors or maternal participants from the ACT clinic
2. Proficient in reading and writing English
3. Cognitively intact such that the study questionnaire can be understood and completed.
4. Participant is willing and able to provide informed consent according to institutional guidelines.

According to institutional and NIH policy, the study will approach and consent research participants regardless of ethnic background.Institutional experience confirms broad representation in this regard.

Exclusion Criteria for acquaintance control group

*Personal history of cancer (for controls aged 18-26 years) or history of having a child diagnosed with cancer (for maternal controls with daughters aged 9-17 years)

A supplemental community control sample (meeting the inclusion and exclusion criteria outlined above) will also be utilized via the subject pool in the Department of Psychology at The University of Memphis.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Maternal participants and young adult females (18-26) enrolled from the ACT clinic will provide contact information for acquaintances in their communities who have daughters (in the young adult arm 18-26 years old peers) roughly the same age as the targeted ACT patient. This will obtain a control sample demographically most like the cancer group. Typically, this will take the form of having the participants access their cell phones, and provide the contact information of the mothers (or 18-26 year old peers) who they identify as potential acquaintance controls. This information will then be used as a means to contact the potential acquaintance control participants. These participants will be mothers with daughters between the ages of 9 and 17 years-of-age or 18-26 year old females. Participants aged 18-26 years will now complete self-reported questionnaires as part of this survey study.
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of HPV vaccination among a large cohort of childhood cancer survivors and an acquaintance control group. | 1 year
To describe the difference in HPV vaccination rate and HPV vaccination intent among preadolescent/adolescent females surviving childhood cancer and an acquaintance control group. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James Klosky, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org